CLINICAL TRIAL: NCT01940575
Title: Clinical Trial to Evaluate the Safety and Efficacy of SkinPlus-Hyal® as Tissue Restorative Biomaterials in the Improvement of Bilateral Nasolabial Fold Wrinkles
Brief Title: Efficacy and Safety Study of SkinPlus-Hyal® to Nasolabial Fold
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: HumanTissueKorea Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-1010-055-001; 06-2013-083 (Other: Seoul National University Bundang Hospital)
Record Dates: First submitted 2013-09-08; First posted 2013-09-12 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Wrinkle
Keywords: Tissue restorative biomaterial; Hyaluronic acid; Restylane®; Wrinkle Severity Rating Scale (WSRS); Global Aesthetic Improvement Scale (GAIS); Nasolabial fold(NLF)

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Restylane® (Active Comparator): Inject Restylane® on right or left nasolabial fold
  Interventions: Device: Restylane®
- SkinPlus-Hyal® (Experimental): Inject SkinPlus-Hyal® on right or left nasolabial fold
  Interventions: Device: SkinPlus-Hyal®

INTERVENTIONS:
Device: SkinPlus-Hyal® — The Injector will administer to the eligible subject the Study Device and Comparator Device (Comparator or Study Device) respectively to the left and right nasolabial fold in a randomized manner.
  Arms: SkinPlus-Hyal®
Device: Restylane® — The Injector will administer to the eligible subject the Study Device and Comparator Device (Comparator or Study Device) respectively to the left and right nasolabial fold in a randomized manner.
  Arms: Restylane®

SUMMARY:
- Study design:Multi-center, randomized, double-masked (Unblinded treating investigators), intra-individual comparison clinical trial

DETAILED DESCRIPTION:
* Subjects:Adults with nasolabial fold
* Investigational Devices:

Study Device: SkinPlus-Hyal® Comparator Device: Restylane®

- Procedure Before Treatment: The subject's eligibility (inclusion/exclusion criteria) will be assessed, and the WSRS of his/her nasolabial fold wil be evaluated by the Investigator Treatment: The Injector will administer to the eligible subject the Study Device and Comparator Device respectively to the left and right nasolabial fold in a randomized manner. Post-Treatment: All subjects will visit the hospital at 2, 8, 16, 24 weeks since the day of administration, and will take pictures of the Nasolabial fold area and undergo efficacy and safety evaluation during each visit. The Photographic evaluator will evaluate the efficacy

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged over 20
2. Subjects who want to correct his/her nasolabial fold and have point 3 or 4 in WSRS of nasolabial fold and visually symmetric
3. Subjects who voluntarily decided the participation of the study and signed the informed consent
4. Subjects who agree contraception

Exclusion Criteria:

1. Subjects who had anaphylaxis or a severe combined allergy, or an allergy to hyaluronic acid
2. Subjects who had eczema, infection, psoriasis, sclerosis, acne on the face
3. Subjects who have a skin disorder on the NLF area
4. Subjects who had permanent implants for dermal augmentation at the NLF area
5. Subjects who had a history of keloid formation or hypertrophic scar
6. Subjects who participated in other clinical trial within 3 months from screening date
7. Female subjects of childbearing potential who disagreed with medically acceptable contraception (e.g., condom, oral contraceptives continuing at least 3 months, injectable or insertable contraceptives, intrauterine contraceptive devices) during the trial
8. Subjects who is Drug abuser or alcoholism
9. Subjects who had previous treatment with Botox within 6 months from screening date
10. Subjects who had previous treatment for wrinkle with Retin-A within 1 months from screening date
11. Subjects who had previous treatment with tissue restorative biomaterials within 18 months from screening date
12. Patients who are not eligible for this study at the medical discretion of the Principal Investigator or Sub-investigator
13. Subjects who had antigen of HIV or type-B Hepatitis
14. Subjects who had anti-coagulant therapy within 2 weeks from the screening date
15. Patients who are not eligible for this study at the medical discretion of the Principal Investigator or Sub-investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2013-07; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
The change in WSRS of the test group and control group | Baseline and 24 weeks
  The change in WSRS of the test group and control group from baseline at 24 weeks as assessed by the Investigator in charge of photographic assessment

SECONDARY OUTCOMES:
The change in WSRS of the test and control groups | baseline and 2, 8, 16, 24 weeks
  The change in WSRS of the test and control groups from baseline at 2, 8, 16, 24 weeks as assessed by the Investigator

OTHER OUTCOMES:
The percentage of subjects whose GAIS is 1 point or above | 2, 8,16, 24 weeks
  The percentage of subjects whose GAIS is 1 point or above at 2, 8, 16, 24 weeks after injection as assessed by the Investigator

CONTACTS AND LOCATIONS:
Overall Officials: Chanyeong - Heo, Ph.D, Principal Investigator — Seoul National University Bundang Hospital
Locations (2):
- South Korea (2):
  - Seoul national university Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Jongno-gu, Seoul